CLINICAL TRIAL: NCT01260259
Title: Effect of Remote Ischemic Preconditioning in Children Undergoing Cardiac Surgery
Brief Title: Seattle Cardiorenal Remote Ischemic Preconditioning Trial
Acronym: SCRIPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Christine Hsu, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CCTR-3953179
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Congenital Heart Disease; Cardiopulmonary Bypass; Myocardial Injury; Acute Kidney Injury; Acute Lung Injury
Keywords: Pediatric; Cardiac; Surgery; Cardiopulmonary; Bypass; Myocardial; Kidney; Lung; Injury
MeSH Terms: conditions — Heart Defects, Congenital; Acute Kidney Injury; Acute Lung Injury; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote Ischemic Preconditioning (RIPC) (Experimental)
  Interventions: Procedure: RIPC
- Control (Sham Comparator)
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: RIPC — RIPC will be elicited in the operating room (OR) after anesthesia induction and before start of surgery. After placement of an arterial line, a tourniquet will be placed over a lower extremity. It will be inflated to 15 mmHg above systolic blood pressure for 5 minutes, and then deflated for 5 minutes. This cycle of inflation-deflation will be repeated another 3 times before surgery.
  Arms: Remote Ischemic Preconditioning (RIPC)
Procedure: Control — In OR, after induction of general anesthesia and arterial line placement, a deflated tourniquet will be placed over the lower extremity for 40 minutes.
  Arms: Control

SUMMARY:
Remote Ischemic Preconditioning (RIPC) is a treatment that may be associated with improved outcomes after cardiac surgery. It can be elicited noninvasively by using a tourniquet to elicit transient ischemia over a lower extremity. It is thought to promote anti-inflammatory and cell survival pathways, and thus protect remote organs against future ischemic injury. We hypothesize that compared to sham treatment, RIPC will be associated with decreased post-operative acute kidney, myocardial, and lung injury.

DETAILED DESCRIPTION:
In children undergoing cardiac surgery and cardiopulmonary bypass (CPB), our primary aims are to determine whether RPC is associated with: 1) decreased AKI and 2) decreased acute myocardial injury. Secondary aims include investigating the effects of RPC on post-procedure: 1)acute lung injury and 2) morbidity/mortality.

ELIGIBILITY:
Inclusion Criteria:

Age birth to 18 years Cardiac surgery with planned cardiopulmonary bypass

Exclusion Criteria:

Any contraindication to compression of lower extremity/extremities Body weight <2 kg Active infection going into surgery On renal replacement therapy (RRT) or mechanical circulatory support going into surgery On inotropic support going into surgery

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2010-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Incidence of acute kidney injury (AKI) | 72 hours
  Serum creatinine (SCr) will be measured at baseline, then on post-operative days 1, 2, and 3.
Incidence of acute myocardial injury | 48 hours
  Troponin-I will be measured at baseline, then 6, 12, 24, and 48 hours post-operative.

SECONDARY OUTCOMES:
Incidence of acute lung injury | 72 hours and duration of hospitalization
  Days on mechanical ventilation, readiness for extubation.
Hospitalization | Duration of post-operative hospitalization
  Number of post-operative days in cardiac intensive care unit (CICU) and hospital.
Mortality | Duration of hospitalization, 30 days post-op, and at last follow-up
Biomarkers for AKI | 72 hours
  Serum and urine will be collected for biomarker discovery.
Inflammation | 72 hours
  Cytokines will be measured at baseline until 72 hours post-operative.

CONTACTS AND LOCATIONS:
Overall Officials: Christine W Hsu, MD, Principal Investigator — Seattle Children's Hospital and University of Washington; Yuk Law, MD, Principal Investigator — Seattle Children's Hospital and University of Washington
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Derived] Law YM, Hsu C, Hingorani SR, Richards M, McMullan DM, Jefferies H, Himmelfarb J, Katz R. Randomized controlled trial of remote ischemic preconditioning in children having cardiac surgery. J Cardiothorac Surg. 2024 Jan 3;19(1):5. doi: 10.1186/s13019-023-02450-8. PMID 38172875